CLINICAL TRIAL: NCT02710019
Title: Back to Reality Series - Harry's Journey: A Video Game About Under Age
Brief Title: Good Shepherd: Back to Reality Series
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Good Shepherd Health Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: McMaster_University
Record Dates: First submitted 2016-02-26; First posted 2016-03-16 (Estimated); Last update posted 2020-11-09 (Actual); Status verified 2018-09

CONDITIONS: Knowledge
Keywords: marijuana use; psychosis; youth; video game
MeSH Terms: conditions — Marijuana Use; Psychotic Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Psychoeducational video games (Experimental): Participants in this group will play the Back to Reality Series video games: (1) Harry's Journey which delivers experiential knowledge about psychosis and marijuana use; (2) Harry's Journal which challenges their understanding of 12 psychiatric symptoms associated with psychosis and (3) the PathwaysToCare Map which uses colourful 3D images and voice-overs to depict actual mental health and addictions services for youth available in Hamilton. These in
  Interventions: Other: Back to Reality Series Video Games
- Control video game (Other): The control video game is a spelling/memory quiz involving with themes from pop culture. The control game will not provide any education about mental health and addictions issues It should be noted that all participants will play both sets of games during their initial and only visit. Participants are randomized to determine which game they will play first during this visit. This is not an RCT or a crossover design. There is no follow up or clinical assessments.
  Interventions: Other: Control Video Game

INTERVENTIONS:
Other: Back to Reality Series Video Games — Back to Reality Series are a psycho-educational video games that provide information about psychosis and marijuana use from the perspective of 'Harry': a character who experiences problems with both issues. The aim is for players to learn how to detect some signs of psychosis and where to seek help for mental health and addictions problems.
  Other Names: Harry's Journal, Harry's Journey, Harry's PathwaysToCare map
  Arms: Psychoeducational video games
Other: Control Video Game — The control video game consists of digital puzzles and spelling game about pop culture. The control games does not have any content related to mental health and addictions problems
  Other Names: Morpheus' Spell
  Arms: Control video game

SUMMARY:
The purpose of this pilot study is to explore whether the Back to Reality series of video games - Harry's Journey, Harry's Journal, and Pathways to care map - increase knowledge of the emotional, social, and psychiatric sequelae of problematic underage marijuana use among homeless and street involved youth. Additional objectives were to explore whether the video games promote awareness of the risk of psychosis associated with regular marijuana use among vulnerable youth.

DETAILED DESCRIPTION:
This project pilots the use of educational video games designed to help youth gain awareness of the risk of mental health issues associated with regular marijuana use. By playing the Back to Reality video games, youths may absorb knowledge about where and how to access community care for symptoms associated with psychosis and problematic cannabis use. The purpose of this study is to pilot test the use of the Back to Reality series at increasing awareness of the social and emotional implications of underage substance use.

This study explores the effects of the Back to Reality video games compared to control video games (no content about mental health and addiction). Street involved and homeless youth registered with Good Shepherd services between the ages of 16 and 19 years of age will be recruited. The results will be assessed using quantitative questionnaires and qualitative interviews. The data will be statistically analyzed for significant differences in knowledge about the risk of psychosis linked to marijuana use among vulnerable youth. The qualitative interview assesses the participants understanding and views of potential emotional, social, and psychiatric sequelae associated with excessive marijuana use during.

ELIGIBILITY:
Inclusion Criteria:

* Homeless or street involved youth
* Registered at any of the Good Shepherd Hamilton Youth programs
* Male, female, or transgender youth from 16-19 years of age as of visit 1.
* Outpatient status
* Each youth must understand the nature this study and sign informed consent

Exclusion Criteria:

* Youth judged by Good Shepherd staff to be at serious suicidal risk.
* Youth who are being discharged from Good Shepherd programming.
* Youth who are currently admitted in an in-patient unit at a hospital.
* Youth who scores 5 or more on the Video Game Playing Problems questionnaire (Teijeiro Salguero & Bersabé-Morán, 2002).
* Youth who do not have the capacity to provide informed consent.

Ages: 16 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2016-05-05 (Actual); Primary Completion 2017-04-18 (Actual); Study Completion 2017-04-18 (Actual)

PRIMARY OUTCOMES:
Psychosis and Cannabis Quiz | 1.5 hour -Post video game playing
  Assess for significant differences in the responses between randomized intervention (Back to Reality series) group versus a control game group with respect to Psychosis and Cannabis Quiz measure. Effect will be tested at a 2-sided α level of 0.05.
Early Psychosis Literacy | 1.5 hour -Post video game playing
  Assess for significant differences in the responses between randomized intervention (Back to Reality series) group versus a control game group with respect to Early Psychosis Literacy measure. Effect will be tested at a 2-sided α level of 0.05.
Video Game Frequency | 1.5 hour -Post video game playing
  Assess for significant differences in the responses between randomized intervention (Back to Reality series) group versus a control game group with respect to Video Game Frequency measure. Effect will be tested at a 2-sided α level of 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Archie, MD, Principal Investigator — McMaster University
Locations (1):
- Good Shepherd, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Roberts MT, Lloyd J, Valimaki M, Ho GW, Freemantle M, Bekefi AZ. Video games for people with schizophrenia. Cochrane Database Syst Rev. 2021 Feb 4;2(2):CD012844. doi: 10.1002/14651858.CD012844.pub2. PMID 33539561